CLINICAL TRIAL: NCT06764342
Title: Adjunctive Effect of Photodynamic Therapy on Halitosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Fernando O Costa, titular professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 30378613.5.0000.5149; NTC02368678 (Registry Identifier: clinicaltrials.gov)
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis; Halitosis
Keywords: halitosis; periodontitis; full-mouth disinfection; antimicrobial photodynamic therapy; real time polymerase chain reaction; bacteria
MeSH Terms: conditions — Periodontitis; Halitosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full-mouth scaling (Active Comparator): Full-mouth ultrasonic and manual periodontal instrumentation
  Interventions: Procedure: full-mouth scaling
- Full-mouth scaling combined with antimicrobial photodynamic therapy (Experimental): Full-mouth ultrasonic and manual periodontal instrumentation combined with antimicrobial photodynamic therapy applied to tongue dorsum and periodontal pockets
  Interventions: Radiation: Full-mouth scaling combined with antimicrobial photodynamic therapy

INTERVENTIONS:
Radiation: Full-mouth scaling combined with antimicrobial photodynamic therapy — After full-mouth scaling procedures antimicrobial photodynamic therapy was carried out using a laser-activated disinfection device with a red laser emission (wavelength: 630 nm, irradiance: 2000-4000 mW/cm², spot size at the probe tip: 8 mm diameter) and high-viscosity methylene blue gel (0.1 mg/mL) which was applied at six spots on the tongue dorsum. Antimicrobial photodynamic therapy was also applied iIn sites with altered periodontal pocket depth (≥ 4mm). The dye remained in the pockets for 10 minutes to ensure full absorption and its excess was rinsed with sterile saline after laser exposure.
  Arms: Full-mouth scaling combined with antimicrobial photodynamic therapy
Procedure: full-mouth scaling — Full-mouth scaling within 24 hours, divided into two sessions of ultrasonic instrumentation followed by manual supra- and subgingival scaling and root planing. Tongue cleaning was performed with a tongue scraper.
  Arms: Full-mouth scaling

SUMMARY:
The present study aims to evaluate bad breath in patients undergoing gingival treatment combined with tongue scraping and laser and to assess its potential benefits for both periodontal and microbiological condition. Firs patients will be selected among those who participated in a privies study. Additional patients will be also invited. They must have gum disease and bad breath. Treatments will be completed within 24 hours and oral samples will be collected with thin paper points. Bad breath will be evaluated by a professional and a specific gas machine.

DETAILED DESCRIPTION:
The present study aims to evaluate halitosis in patients undergoing non-surgical periodontal therapy [(Full-mouth disinfection (FMD) combined with tongue scraping and antimicrobial photodynamic therapy (aPDT), and to assess its potential benefits for both periodontal and microbiological condition. A pilot study will be performed with participants who took part almost 10 years ago in the study NCT02368678. They will be invited by phone contact. In addition, new participants will be recruited by convenience in dental clinics from the Federal University of Minas Gerais until completion of 20 participants per group. Individuals with stage III periodontitis and halitosis (organoleptic method > 2), will be allocated into two periodontal treatment groups. Halitosis will be assessed using the organoleptic method and gas chromatography (OralChroma device) at three time points: before and after treatments. Microbiological samples will be collected before and after treatments from periodontal pockets and pooled samples from the tongue dorsum. These samples will be analyzed by using real-time PCR (q-PCR) aiming at detecting target bacterial species.

ELIGIBILITY:
Inclusion Criteria:

* self-reported halitosis;
* organoleptic score >2;
* stage III periodontitis;
* at least 14 teeth.

Exclusion Criteria:

* smokers or former smokers;
* individuals diagnosed with diabetes and/or immune diseases;
* pregnant or lactating women;
* individuals with removable partial dentures and/or fixed or removable orthodontic appliances;
* systemic use of antibiotics or anti-inflammatory drugs in the last three months; - individuals who required prophylactic antibiotics for periodontal exams and treatments;
* individuals who regularly used or had used any type of mouthwash in the past three months;
* individuals who underwent periodontal treatment in the six months prior to the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
sulfur volatile compounds changes | baseline versus 21 and 45 days after treatment
  pre and post-treatment changes in levels (parts per billion) of CH3SH, a sulfur volatile compound

SECONDARY OUTCOMES:
Changes in periodontal probing depth | baseline versus 45 days after treatment
  Pre and pos-treatment changes in periodontal pocket depth (mm)
Changes in organoleptic testing | Baseline versus 45 days after treatment
  Pre and post-treatment changes in organoleptic scores
Changes in tongue total bacteria count | baseline versus 45 days after treatment
  Pre- and post-treatment changes in total bacteria counts from tongue dorsal samples

CONTACTS AND LOCATIONS:
Overall Officials: Fernando O Costa, doctorate, Principal Investigator — Federal University of Minas Gerais, Dental School
Locations (1):
- Federal University of Minas Gerais, Dental School, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No
Data will be analyzed by group and using numerical codes avoiding individual personal data identification. Data access will be protected by password.